CLINICAL TRIAL: NCT06886269
Title: A Phase 1, Open-label, Mass Balance Study to Investigate the Absorption, Distribution, Metabolism, and Excretion of 14C-VX-993 Following Single Oral Administration in Healthy Subjects
Brief Title: A Study to Evaluate How the Body Processes 14C-VX-993 After a Single Oral Dose
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Vertex Pharmaceuticals Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VX24-993-007
Record Dates: First submitted 2025-03-14; First posted 2025-03-20 (Actual); Last update posted 2025-06-18 (Actual); Status verified 2025-06

CONDITIONS: Pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- 14C VX-993 (Experimental): Participants will receive a single oral dose of 14C-VX-993 after an overnight fast of at least 8 hours.
  Interventions: Drug: 14C-VX-993

INTERVENTIONS:
Drug: 14C-VX-993 — Solution for Oral Administration.

SUMMARY:
The purpose of the study is to evaluate the routes and rate of elimination and recovery of total radioactivity (TRA) and characterize the Pharmacokinetic (PK) of VX-993 after a single oral dose of 14C-VX-993.

DETAILED DESCRIPTION:
This clinical trial information was submitted voluntarily under the applicable law and, therefore, certain submission deadlines may not apply. (That is, clinical trial information for this applicable clinical trial was submitted under section 402(j)(4)(A) of the Public Health Service Act and 42 CFR 11.60 and is not subject to the deadlines established by sections 402(j)(2) and (3) of the Public Health Service Act or 42 CFR 11.24 and 11.44.)

ELIGIBILITY:
Key Inclusion Criteria:

* Body mass index (BMI) of 18.0 to 32.0 kilogram per meter square (kg/m^2), inclusive
* A total body weight of more than (>) 50 kg
* Participants must have at least 1 regular bowel movement per day

Key Exclusion Criteria:

* History of febrile illness or other acute illness that has not fully resolved within 14 days before the first dose of study drug
* Any condition possibly affecting drug absorption, distribution, metabolism, or excretion
* Exposure to any non-environmental radiation within 12 months of dosing
* Participation in more than 1 radiolabeled study (if prior radiation exposure unknown) or participation in more than 3 radiolabeled studies (if radiation exposure known) in the 12 months before dosing or if the annual whole body radiation exposure from previous studies (including this dosing) exceeds FDA-allowed maximum whole body radiation exposure of 5000 mrem

Other protocol defined Inclusion/Exclusion criteria may apply.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2025-03-21 (Actual); Primary Completion 2025-05-17 (Actual); Study Completion 2025-05-17 (Actual)

PRIMARY OUTCOMES:
Terminal Phase Rate Constant (λz) of VX-993 in Plasma | From Day 1 up to Day 25
Area Under the Concentration Versus Time Curve From the Time of Dosing to the Last Measurable Concentration (AUC0-tlast) of VX-993 in Plasma | From Day 1 up to Day 25
Area Under the Concentration Versus Time Curve From the Time of Dosing Extrapolated to Infinity (AUC0-inf) of VX-993 in Plasma | From Day 1 up to Day 25
Apparent Clearance (CL/F) of VX-993 in Plasma | From Day 1 up to Day 25
Maximum Observed Plasma Concentration (Cmax) of VX-993 in Plasma | From Day 1 up to Day 25
Time for VX-993 to Reach Maximum Concentration (Tmax) in Plasma | From Day 1 up to Day 25
Apparent Volume of Distribution (Vz/F) (Based on the Terminal Phase) of VX-993 in Plasma | From Day 1 up to Day 25
Terminal Phase Rate Constant (λz) of Total Radioactivity (TRA) in Whole blood and Plasma | From Day 1 up to Day 25
Amount of Radioactivity Excreted (Ae) of TRA in Urine, Feces and Vomitus (if applicable) | Pre dose up to Day 25
AUC0-tlast of TRA in Whole blood and Plasma | From Day 1 up to Day 25
AUC0-inf of TRA in Whole blood and Plasma | From Day 1 up to Day 25
CL/F of TRA in Whole blood and Plasma | From Day 1 up to Day 25
Renal Clearance (CLr) of TRA in Urine and Feces | Pre dose up to Day 25
Cmax of TRA in Whole blood and Plasma | From Day 1 up to Day 25
Fraction (percent) of Dose Excreted Unchanged in Urine of TRA | Pre dose up to Day 25
Tmax of TRA in Whole blood and Plasma | From Day 1 up to Day 25
Apparent Volume of Distribution (Based on the Terminal Phase) of TRA in Whole blood and Plasma | From Day 1 up to Day 25
Amount of VX-993 and Metabolites, Expressed as a percent of TRA, in Plasma, Urine and Feces | From Day 1 up to Day 25

SECONDARY OUTCOMES:
Metabolite Profiling and Identification in Plasma, Urine, and Feces | From Day 1 up to Day 25
Terminal Phase Rate Constant (λz) of VX-993 Metabolites in Plasma and Urine (if applicable) | From Day 1 up to Day 25
Amount of radioactivity excreted (Ae) of VX-993 Metabolites in Urine and Feces | Pre dose up to Day 25
AUC0-last of VX-993 Metabolites in Plasma | From Day 1 up to Day 25
AUC0-inf of VX-993 Metabolites in Plasma | From Day 1 up to Day 25
CL/F of VX-993 Metabolites in Plasma | From Day 1 up to Day 25
CLr of VX-993 Metabolites in Urine | From Day 1 up to Day 25
Cmax of VX-993 Metabolites in Plasma | From Day 1 up to Day 25
Fraction (percent) of Dose Excreted Unchanged in Urine of VX-993 Metabolites | Pre dose up to Day 25
Tmax of VX-993 Metabolites in Plasma | Day 1 up to Day 25
Apparent Volume of Distribution (Based on the Terminal Phase) of VX-993 Metabolites in Plasma | Day 1 up to Day 25
Safety and Tolerability as Assessed by Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs) | Day 1 up to Day 35
Safety and Tolerability as Assessed by Number of Participants With Clinically Meaningful Findings in Columbia Suicide Severity Rating Scale (C-SSRS) Responses | Pre-dose up to Day 35

CONTACTS AND LOCATIONS:
Locations (1):
- Celerion - Lincoln, Lincoln, Nebraska, United States

IPD SHARING:
Plan to Share IPD: No
Details on Vertex data sharing criteria and process for requesting access can be found at: https://www.vrtx.com/independent-research/clinical-trial-data-sharing